CLINICAL TRIAL: NCT02071108
Title: Safety and Performance Study of the Shockwave Lithoplasty System
Acronym: DISRUPT-PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD 0083
Record Dates: First submitted 2014-02-22; First posted 2014-02-25 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithoplasty Treatment (Experimental): Shockwave Lithoplasty System
  Interventions: Device: Shockwave Lithoplasty System

INTERVENTIONS:
Device: Shockwave Lithoplasty System

SUMMARY:
To study the safety and performance of the Shockwave Medical Lithoplasty System in subjects to demonstrate that the Shockwave device can safely and effectively deliver localized shockwave energy for balloon dilatation of calcified, stenotic, infrainguinal peripheral arteries.

DETAILED DESCRIPTION:
Shockwave Medical, Inc. intends to conduct a prospective, single-arm, multi-center, clinical study designed to evaluate the safety and performance of the Shockwave Lithoplasty System in subjects with moderate to heavily calcified peripheral arteries with 3.50mm to 7.0mm reference vessel diameter at the target site. The Shockwave Lithoplasty System is indicated to generate sonic shockwave energy within the target treatment site and disrupt calcium within the lesion to allow for subsequent dilation of a peripheral artery stenosis using low balloon pressure. Up to thirty-five (35) subjects will be enrolled and treated with Lithoplasty to yield thirty (30) evaluable subjects complete the study assuming a 15% lost to follow-up rate.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to comply with all assessments in the study.
2. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
3. Age of subject is >18.
4. Rutherford Clinical Category 2, 3, or 4.
5. Resting ankle-brachial index (ABI) of ≤0.90, or ≤0.75 after exercise, of the target leg.
6. Moderate to severe calcification of target lesion(s) per pre-procedure CT scan. (Calcification must be: 1) ≥180 degrees circumferential at some point in the lesion and 2) extend ≥50 percent length of lesion or absolute length ≥20mm.)
7. Estimated life expectancy >1 year.

Exclusion Criteria:

1. Rutherford Clinical Category 5 and 6.
2. Subject has active infection in the target leg.
3. Planned major amputation of the target leg (transmetatarsal or higher).
4. In-stent restenosis within the target lesion(s).
5. Highly tortuous arteries (bends greater than 30 degrees over the arc length of the balloon).
6. Chronic total occlusion of the target lesion(s).
7. Target lesion(s) within native or synthetic vessel grafts.
8. Chronic total occlusion of inflow vessel.
9. Lesion in contralateral limb requiring intervention within the next 30 days.
10. History of prior endovascular or surgical procedure on the index limb within the past 30 days.
11. Subject has significant stenosis (>50% stenosis) or occlusion of inflow tract (upstream disease) not successfully treated with plain old balloon angioplasty or stent and without complications before target lesion(s) treatment.
12. Subject requires treatment of a peripheral lesion on the ipsilateral limb distal to the target lesion(s) at the time of the enrollment / index procedure.
13. Subject has a known coagulopathy or has a bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter, or international normalized ratio >1.5.
14. Subject in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated.
15. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
16. Subject has known allergy to urethane, nylon, or silicone.
17. Myocardial infarction within 60 days prior to enrollment.
18. History of stroke within 60 days prior to enrollment.
19. History of unstable coronary artery disease or other uncontrollable comorbidity resulting in hospitalization within the last 60 days prior to enrollment.
20. History of thrombolytic therapy within two weeks of enrollment.
21. Subject has acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L), or on dialysis.
22. Subject is pregnant or nursing.
23. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
24. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Bad Krozingen; Andrew Holden, MD, Principal Investigator — Auckland City Hospital
Locations (3):
- Medizinische Universitaet Graz, Graz, Graz, Austria
- Department of Angiology - Universitats Herzzentrum Freiburg, Bad Krozingen, Baden-Wurttemberg, Germany
- Auckland City Hospital, Auckland, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three investigational sites in Austria and New Zealand participated in the study. Between January 2014 and September 2014, a total of 35 subjects and 39 lesions of the superficial femoral and popliteal arteries were enrolled in the Full Analysis Cohort of the study and treated with the investigational device.
Groups:
- Lithoplasty Treatment: All subjects were treated with the Shockwave Medical Peripheral Lithoplasty System
Period: Overall Study
Arm/Group | Lithoplasty Treatment
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Lithoplasty Treatment: Shockwave Medical Peripheral Lithoplasty System
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 29
Region of Enrollment [Number; unit: participants]
  New Zealand | 7
  Austria | 28

OUTCOME MEASURES:

1. Primary Outcome: Composite of New-onset Major Adverse Events (MAE)
Description: Need for emergency surgical revascularization of target limb. Unplanned target limb amputation (above the ankle). Symptomatic thrombus or distal emboli, defined as clinical signs or symptoms of thrombus or distal emboli detected in the treated limb in the area of the treated lesion, or distal to the treated lesion, after the index procedure or noted angiographically, and requiring mechanical or pharmacologic means to improve flow. Perforations and dissections of grade D or greater that require an intervention to resolve, including bail-out stenting.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
participants | 0

2. Primary Outcome: Procedural Success:
Description: The ability of the Shockwave Medical Lithoplasty System to achieve a post-Shockwave residual diameter stenosis of <50% (with or without adjunctive Percutaneous Transluminal Angioplasty therapy) as assessed by quantitative angiography via core lab evaluation.
Time Frame: Day of Procedure
Population: Full Analysis Cohort - All subjects who were enrolled in the study and where delivery of the Shockwave Medical Peripheral Lithoplasty treatment was attempted.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Number analyzed (lesions) | 39
percentage of lesions | 100 [91.0 to 100.0]

3. Secondary Outcome: Device Success
Description: The ability of the Shockwave Medical Lithoplasty System to achieve a post-Shockwave residual diameter stenosis of <50% (without adjunctive percutaneous transluminal angioplasty therapy) as assessed via quantitative angiography via core lab evaluation.
Time Frame: Day of Procedure
Population: Full Analysis Cohort - All subjects who were enrolled in the study and where delivery of the Shockwave Medical Peripheral Lithoplasty treatment attempted
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Number analyzed (lesions) | 39
percentage of lesions | 87.2 [72.6 to 95.7]

4. Secondary Outcome: Clinical Success:
Description: The ability of the Shockwave Medical Lithoplasty System to achieve a post-Shockwave residual diameter stenosis of <50% (with or without adjunctive percutaneous transluminal angioplasty therapy) as assessed by the investigator via visual estimate and freedom from procedural major adverse events.
Time Frame: Day of Procedure
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
percentage of participants | 100 [90.0 to 100.0]

5. Secondary Outcome: Technical Success:
Description: The ability of the Shockwave Medical Lithoplasty System to delivery ShockWave treatment to the desired location in the target vessel. Up to two Shockwave Medical Lithoplasty Systems maybe used to complete treatment in the target vessel.
Time Frame: Day of Procedure
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Number analyzed (lesions) | 39
percentage of lesions | 97.4 [86.5 to 99.9]

6. Secondary Outcome: Freedom From Major Adverse Events
Description: Freedom from Major Adverse Events at 30 days.
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
percentage of participants | 100

7. Secondary Outcome: Freedom From Target Lesion Revascularization (TLR)
Description: Freedom from Target Lesion Revascularization (TLR) at 30 days
Time Frame: 30 days
Population: Per-Protocol Cohort - the group of subjects who were enrolled in the study and where delivery of the Shockwave Medical Peripheral Lithoplasty treatment was successfully completed
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Number analyzed (lesions) | 39
percentage of lesions | 100

8. Secondary Outcome: Patency
Description: Vessel patency at 30 days by Doppler Ultrasound defined as freedom from greater than 50% restenosis (as assessed by Duplex ultrasound peak systolic velocity ratio of ≥2.5).
Time Frame: 30 days
Population: Full Analysis Cohort - All subjects who were enrolled in the study and where delivery of the Shockwave Medical Peripheral Lithoplasty treatment was attempted. Due to device malfunctions, one subject received partial treatment. To provide a more accurate account of actual device usage, the subject was omitted from the analysis of device usage only.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 34
Number analyzed (lesions) | 38
percentage of lesions | 100 [90.7 to 100.0]

9. Secondary Outcome: Ankle Brachial Index (ABI)
Description: Change in Ankle Brachial Index (ABI) of the target limb at 30 days. The Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm.
Time Frame: Baseline and 30 days
Population: Per-Protocol Cohort - the group of subjects who were enrolled in the study and where delivery of the Shockwave Medical Peripheral Lithoplasty treatment was successfully completed. Four subjects were not included in the analysis because ABI could not be measured due to non-compressible disease that inhibited accurate ABI measurement.
Measure: Mean (95% Confidence Interval); unit: change in ABI score from baseline
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 31
change in ABI score from baseline | 0.3 [0.2 to 0.4]

10. Secondary Outcome: Rutherford Clinical Category
Description: Change in Rutherford Clinical Category (RCC) at 30 days. RCC identifies three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss. Grade I includes Category 0 - Asymptomatic, Category 1 - Mild claudication, Category 2 - Moderate claudication, and Category 3 - Severe claudication. Grade II includes Category 4 - Ischemic rest pain and Category 5 - Minor tissue loss. Grade III includes Category 6 - Ulceration or grangrene. Change of at least 2 categories considered statistically significant.
Time Frame: Baseline and 30 days
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: change in RCC from baseline
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
change in RCC from baseline | -2.5 [-2.7 to -2.2]

11. Secondary Outcome: Freedom From Major Adverse Events
Description: Freedom from Major Adverse Events at 6 months
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
percentage of participants | 100

12. Secondary Outcome: Freedom From Target Lesion Revascularization (TLR)
Description: Freedom from Target Lesion Revascularization (TLR) at 6 months
Time Frame: 6 months
Population: as for outcome 7
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Number analyzed (lesions) | 39
percentage of lesions | 100

13. Secondary Outcome: Patency
Description: Vessel patency at 6 months at Doppler Ultrasound defined as freedom from greater than 50% restenosis (as assessed by Duplex ultrasound peak systolic velocity ratio of =2.5).
Time Frame: 6 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Number analyzed (lesions) | 39
percentage of lesions | 82.1 [66.5 to 92.5]

14. Secondary Outcome: Ankle Brachial Index (ABI)
Description: Change in Ankle Brachial Index (ABI) of the target limb at 6 months. The Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm.
Time Frame: Baseline and 6 months
Population: Per-Protocol Cohort - the group of subjects who were enrolled in the study and where delivery of the Shockwave Medical Lithoplasty treatment was successfully completed
Measure: Mean (95% Confidence Interval); unit: Ankle Brachial Index
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 31
Ankle Brachial Index | 1.0 [0.9 to 1.1]

15. Secondary Outcome: Rutherford Clinical Category
Description: Change in Rutherford Clinical Category (RCC) at 6 months. RCC identifies three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss. Grade I includes Category 0 - Asymptomatic, Category 1 - Mild claudication, Category 2 - Moderate claudication, and Category 3 - Severe claudication. Grade II includes Category 4 - Ischemic rest pain and Category 5 - Minor tissue loss. Grade III includes Category 6 - Ulceration or grangrene. Change of at least 2 categories considered statistically significant.
Time Frame: Baseline and 6 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: Rutherford Clinical Category
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Rutherford Clinical Category | 0.4 [0.2 to 0.6]

16. Other Pre Specified Outcome: Exploratory Endpoint
Description: The clinical protocol provided for an Exploratory Secondary Endpoint to assess the ability of the device to achieve ≤30% residual stenosis without adjunctive PTA as assessed by the investigator via visual estimate.
Time Frame: Day of Procedure
Population: as for outcome 7
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Lithoplasty Treatment
Number analyzed (Participants) | 35
Number analyzed (lesions) | 39
percentage of lesions | 87

ADVERSE EVENTS:
Time Frame: through 30 days and 6 months
Arm/Group | Lithoplasty Treatment
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithoplasty Treatment (N=35)
Need for emergency surgical revascularization of target limb (Surgical and medical procedures) | 0 (0)
Unplanned target limb amputation (above the ankle) (Surgical and medical procedures) | 0 (0)
Symptomatic thrombus or distal emboli (Injury, poisoning and procedural complications) | 0 (0) — clinical signs or symptoms of thrombus or distal emboli detected in treated limb in area of treated lesion or distal to treated lesion after index procedure or noted angiographically and requiring mechanica or pharmacological means to improve flow
Perforations and dissections of grade D or greater that require an intervention to resolve (Injury, poisoning and procedural complications) | 0 (0) — includes bail-out stenting
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithoplasty Treatment (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Photokeratitis (Eye disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Vessel puncture site haematoma (General disorders) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Endarterectomy (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No